CLINICAL TRIAL: NCT04701671
Title: Executive Functioning, Weight Trajectories, and Loss of Control Eating in Children With Overweight/Obesity: A Prospective Study
Brief Title: Project THINK: Trajectories of Health, Ingestive Behaviors, and Neurocognition in Kids
Status: Recruiting | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: Brown University (Other); The Miriam Hospital (Other); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Andrea Goldschmidt, Associate Professor, University of Pittsburgh
Other Study IDs: STUDY21070033; R01DK120597 (NIH)
Record Dates: First submitted 2021-01-06; First posted 2021-01-08 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Pediatric Obesity; Binge-Eating Disorder
Keywords: Loss of Control Eating; Executive Functioning; Pubertal Development
MeSH Terms: conditions — Pediatric Obesity; Binge-Eating Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (6):
- Normal Weight Control, no MRI-scan (30 participants): Adolescents with a BMI percentile under 85% who are not randomly assigned to undergo MRI scans at baseline and 18-months.
  Interventions: Behavioral: Observational (not including MRI scanning)
- Normal Weight Control with MRI-scan (30 participants): Adolescents with a BMI percentile under 85% who are randomly assigned to undergo MRI scans at baseline and 18-months.
  Interventions: Behavioral: Observational (including MRI scanning)
- Overweight Control, no MRI-scan (30 participants): Adolescents with a BMI percentile at 85% or higher who are not randomly assigned to undergo MRI scans at baseline and 18-months.
  Interventions: Behavioral: Observational (not including MRI scanning)
- Overweight Control with MRI-scan (30 participants): Adolescents with a BMI percentile at 85% or higher who are randomly assigned to undergo MRI scans at baseline and 18-months.
  Interventions: Behavioral: Observational (including MRI scanning)
- Overweight/Obese Experimental, no MRI-scan (30 participants): Adolescents with a BMI percentile at 85% or higher, who report loss of control eating episodes and are not randomly assigned to undergo MRI scans at baseline and 18-months.
  Interventions: Behavioral: Observational (not including MRI scanning)
- Overweight/Obese Experimental with MRI-scan (30 participants): Adolescents with a BMI percentile at 85% or higher, who report loss of control eating episodes and are randomly assigned to undergo MRI scans at baseline and 18-months.
  Interventions: Behavioral: Observational (including MRI scanning)

INTERVENTIONS:
Behavioral: Observational (not including MRI scanning) — Observational data will be obtained through self-report measures, parental report measures, cognitive assessments, and a semi-structured interview.
  Groups: Normal Weight Control, no MRI-scan (30 participants); Overweight Control, no MRI-scan (30 participants); Overweight/Obese Experimental, no MRI-scan (30 participants)
Behavioral: Observational (including MRI scanning) — Observational data will be obtained through self-report measures, parental report measures, cognitive assessments, fMRI imaging, and a semi-structured interview.
  Groups: Normal Weight Control with MRI-scan (30 participants); Overweight Control with MRI-scan (30 participants); Overweight/Obese Experimental with MRI-scan (30 participants)

SUMMARY:
Overweight/obesity and loss of control eating (characterized by the sense that one cannot control what or how much one is eating) are prevalent among children and adolescents, and both are associated with serious medical and psychosocial health complications. Although our recently published data suggest that youth with these conditions may have relative deficits in neurocognitive functioning, particularly working memory, understanding of how these processes and their neural correlates are related to change and stability in eating and weight-related outcomes over time is limited, thereby impeding development of targeted, optimally timed interventions. The present study aims to assess prospective associations between general and food-specific executive functioning and underlying neural substrates, and eating and weight outcomes among children at varying levels of risk overweight/obesity and eating disorders, which will help guide research efforts towards the development of effective prevention and intervention strategies.

DETAILED DESCRIPTION:
The current study will examine prospective associations among general and food-specific EF and related neural substrates, and the developmental course of weight gain and LOC eating from middle childhood through early adolescence. Specific aims are to:

1. Investigate prospective associations between general and food-specific EF and z-BMI trajectories. We expect that across risk groups, a) poorer baseline performance on both general and food-specific behavioral EF measures will predict steeper z-BMI gain trajectories; and b) worsening general and food-specific EF will track with the steepest z-BMI gain trajectories.
2. Investigate associations between general and food-specific EF and LOC eating trajectories. We expect that across risk groups, a) poorer baseline performance on general and food-specific behavioral EF measures will predict worsening course of LOC eating; and b) worsening general and food-specific EF will track with worsening course of LOC eating.
3. Investigate prospective associations between EF neural substrates and trajectories of z-BMI and LOC eating. We expect that across risk groups, a) greater activation in prefrontal regions associated with EF (e.g., dorsolateral prefrontal cortex, dorsal cingulate, parietal cortex) during general and food-specific WM tasks, and b) smaller decreases in activation of these regions over 18 months, will predict steeper z-BMI gain trajectories and worsening course of LOC eating.

ELIGIBILITY:
Inclusion Criteria:

* Not currently taking any medications known to affect weight or appetite
* Free of any current or past medical or psychiatric conditions known to significantly affect eating or weight (e.g., diabetes, bulimia nervosa), with the exception of binge eating disorder
* In the low average range or higher on measures of general intellectual functioning
* Free of any conditions affecting executive functioning (e.g., recent concussion, history of traumatic brain injury)
* Fluent in English, and able to read and comprehend study materials
* Not currently pregnant

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Participants will include 180 children (9-12y) representing a spectrum of risk for eating and weight disorders, including overweight/obese (BMI ≥ 85th age- and sex-adjusted percentile) with LOC eating (n=60), overweight/obese without LOC eating (n=60), and healthy weight without LOC eating (5th percentile ≤ BMI < 85th percentile; n=60).
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2020-12-10 (Actual); Primary Completion 2028-05-09 (Estimated); Study Completion 2028-05-09 (Estimated)

PRIMARY OUTCOMES:
BMI (Body Mass Index) | Change in BMI from baseline to 24 months
  BMI will be assessed using height and weight (cm/g)
Eating Behavior | Change in eating behavior from baseline to 24 months
  Eating behavior will be assessed using the Eating Disorder Examination (EDE), a semi-structured interview. Global scores are calculated, with higher scores indicating higher disordered eating symptomology.
General Executive Functioning | Change in general executive functioning from baseline to 24 months
  A general n-back task that will involve continuous presentation of neutral stimuli (letters or numbers). Participants indicate via button press whether the target (current) stimulus was presented n items ago.
Food-Specific Executive Functioning | Change in food-specific executive functioning from baseline to 24 months
  A food-specific WM task that involves continuous presentation of stimuli representing food and non-food items. Participants indicate via button press whether the target (current) stimulus was presented n items ago.

CONTACTS AND LOCATIONS:
Overall Officials: Andrea B. Goldschmidt, Ph.D., Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - University of PIttsburgh, Pittsburgh, Pennsylvania
  - Weight Control & Diabetes Research Center, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2022-11-04): https://cdn.clinicaltrials.gov/large-docs/71/NCT04701671/ICF_002.pdf